CLINICAL TRIAL: NCT02069379
Title: Endogenous Opioid Activity and Affective State in Insulin Resistant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alison Berent-Spillson, Research Investigator, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HUM00066696; K01MH095920 (NIH)
Record Dates: First submitted 2013-11-06; First posted 2014-02-24 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Depression; Insulin Resistance; Metabolic Syndrome
Keywords: Metabolic syndrome; Insulin resistance; Mu-opioid system; Depression; Emotion regulation
MeSH Terms: conditions — Depression; Insulin Resistance; Metabolic Syndrome; Emotional Regulation | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Controls (No Intervention): metabolically healthy controls will participate in baseline assessments only, and will not be randomized to the placebo and metformin treatment arms.
- Metformin (Experimental): 16 weeks treatment with metformin (insulin sensitizing treatment)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo comparator to metformin treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Women classified as insulin resistant will participate in both a placebo and a metformin treatment arm, each lasting about 16 weeks. Women will be randomized to order of treatment arms.
  Other Names: Glucophage; Glumetza; Fortamet; Riomet
  Arms: Metformin
Drug: Placebo — Placebo capsules prepared identically to Metformin capsules
  Other Names: Sugar pills
  Arms: Placebo

SUMMARY:
Insulin resistance, a primary component of the metabolic syndrome, is an escalating phenomenon in the United States, and confers an increased risk of depression and mood disorder, particularly in women. The relationship between metabolic and mood disorders may be mediated by endogenous opioid activity in limbic brain regions. We propose to examine affective state and μ- opioid system function in insulin resistant women, and change in response to insulin sensitizing treatment, through the following specific aims and hypotheses:

Establish relationship between insulin resistance, affective state, and μ-opioid receptor function.

1. Insulin resistant women will have greater μ-opioid receptor availability at baseline, and a larger response to stress challenge than non-insulin resistant women
2. Insulin resistant women will have greater negative affective state at baseline, and a greater emotional response to stress challenge than non-insulin resistant women.
3. Mediational analyses will reveal that the relationship between insulin resistance and negative affect is mediated by μ-opioid receptor function and neural activation in the amygdala and nucleus accumbens affect-regulating regions.

Examine effects of insulin regulation on μ-opioid receptor function and affective state.

1. Improved insulin sensitivity will be accompanied by decreased μ-opioid receptor availability at baseline and a reduced response to stress challenge. Degree of change in baseline receptor availability and response to stress challenge after treatment will correlate with degree of insulin regulation.
2. Improved insulin sensitivity will be associated with improved affective state at baseline, and with a reduced emotional response to stress challenge. Degree of change in affective state and emotional response to stress challenge after treatment will correlate with degree of insulin regulation.
3. Mediational analyses will reveal that the change in affective state after insulin regulation is mediated by change in μ-opioid receptor function and neural activation in the amygdala and nucleus accumbens.

The expected results would suggest a role for the endogenous μ-opioid system in mediating the relationship between metabolic function and emotional processes.

DETAILED DESCRIPTION:
The objective of this study is to examine the role of the endogenous mu-opioid system in mediating the relationship between metabolic dysfunction and depressive symptoms in reproductive aged women.

PET image data was unable to be analyzed due to PET equipment replacement midway through study, leaving PET images collected at beginning of study incompatible with PET images collected later in study.

Due to insufficient enrollment in treatment arms, the 20 or 40 week data was unusable for analytic goals, so the study was re-framed for what could usefully be learned about baseline characteristics among the study populations and the originally planned outcome measures were amended to only to those that related to understanding the baseline population.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18-40 years old
* metabolically healthy or insulin resistant (insulin sensitivity > 1.89x10-4 (min-1 x µU-1 x mL-1; calculated by minimal model assessment of glucose tolerance test)
* body mass index (BMI = weight (kg) / height2 (m2)) between 18 kg/m2 and 35 kg/m2.
* Women with mild or moderate depressive symptoms not meeting the criteria for Major Depressive Disorder will be included.

Exclusion Criteria:

* men
* left handed
* acute medical illness
* uncorrected thyroid disease
* diabetes (fasting glucose ≥126 mg/dL)\
* neurological disease
* major depression
* substance abuse
* MRI contraindications (claustrophobia, pacemakers, pumps, metallic agents or devices)
* severe calorie restriction
* intense physical exercise ≥1 hour/day
* smoking within 6 months
* hormonal, insulin sensitizing, or centrally acting medications within 2 months
* pregnancy within 6 months
* lactation
* cardiac or pulmonary insufficiency
* liver or renal insufficiency (>2.5 x normal transaminases levels, plasma creatinine ≥1.4 mg/dL)
* history of lactic acidosis
* BMI ≥35 kg/m2
* opioid allergy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Berent-Spillson, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical School, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Resistant Participants (Placebo First): Women classified as insulin resistant will participate in both a placebo and a metformin treatment arm, each lasting about 16 weeks. Women will be randomized to order of treatment arms.
- Insulin Resistant Participants (Metformin First): Women classified as insulin resistant and randomized to Metformin treatment arm 1st and Placebo treatment arm 2nd
- Insulin Resistant (Not Randomized): Insulin resistant participants not randomized to treatment arms
Period: Baseline Measurements
Arm/Group | Controls | Insulin Resistant Participants (Placebo First) | Insulin Resistant Participants (Metformin First) | Insulin Resistant (Not Randomized)
Started | 30 | 4 | 2 | 6
Baseline Measurements Taken | 30 | 4 | 2 | 6
Completed | 27 | 4 | 2 | 4
Not Completed | 3 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Ineligible based on initial assessments | 2 | 0 | 0 | 2
Period: First Treatment Arm
Arm/Group | Controls | Insulin Resistant Participants (Placebo First) | Insulin Resistant Participants (Metformin First) | Insulin Resistant (Not Randomized)
Started | 0 (Controls are not involved after initial baseline collection) | 4 | 2 | 0 (Insulin resistant woman not randomized are not involved after initial baseline collection)
Completed | 0 | 3 | 1 | 0
Not Completed | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Period: Washout Period (4 Weeks)
Arm/Group | Controls | Insulin Resistant Participants (Placebo First) | Insulin Resistant Participants (Metformin First) | Insulin Resistant (Not Randomized)
Started | 0 (Controls are not involved after initial baseline collection) | 3 | 1 | 0 (Insulin resistant woman who were not randomized are not involved after initial baseline collection)
Completed | 0 | 1 | 1 | 0
Not Completed | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Unrelated event | 0 | 1 | 0 | 0
Period: Second Treatment Arm
Arm/Group | Controls | Insulin Resistant Participants (Placebo First) | Insulin Resistant Participants (Metformin First) | Insulin Resistant (Not Randomized)
Started | 0 (Controls are not involved after initial baseline collection) | 1 | 1 | 0 (Insulin resistant women who are not randomized are not involved after initial baseline collection)
Completed | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All insulin resistant women are grouped together for baseline characteristics, as these measurements were taken prior to treatment arm randomization
Groups:
- Insulin Resistant Participants: Women classified as insulin resistant will participate in both a placebo and a metformin treatment arm, each lasting about 16 weeks. Women will be randomized to order of treatment arms.
- Total: Total of all reporting groups
Arm/Group | Controls | Insulin Resistant Participants | Total
Number analyzed (Participants) | 30 | 12 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 12 | 42
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 12 | 42
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 30 | 12 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 13 | 7 | 20
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 12 | 42
Glucose [Mean (Standard Deviation); unit: mg/dL] | 80.29 (5.33) | 84.67 (9.99) | 81.60 (7.21)
Plasma Insulin Levels [Mean (Standard Deviation); unit: mIU/L] | 10.18 (1.99) | 18.61 (3.36) | 12.71 (4.61)
HOMA Insulin Resistance (IR) [Mean (Standard Deviation); unit: HOMA IR] | 2.01 (0.42) | 3.94 (1.11) | 2.56 (1.12)

OUTCOME MEASURES:

1. Primary Outcome: Mu-opioid Receptor Binding Potential in Left Nucleus Accumbens, Resting State
Description: Mu-opioid neurotransmission in limbic brain regions at baseline and change from baseline after metformin treatment
Time Frame: Baseline, 20 weeks, 40 weeks
Population: PET scanners available were replaced for other institutional reasons which resulted in image production so incompatible as to be not comparable. Therefore PET image data files were unable to be analyzed due to inconsistencies with imaging techniques.
Arm/Group | Controls | Metformin | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Mu-opioid Receptor Binding Potential in Right Nucleus Accumbens, Resting State
Description: Mu-opioid neurotransmission in limbic brain regions at baseline and change from baseline after metformin treatment
Time Frame: Baseline, 20 weeks, 40 weeks
Population: as for outcome 1
Arm/Group | Controls | Metformin | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Mu-opioid Receptor Binding Potential in Left Amygdala, Resting State
Description: Mu-opioid neurotransmission in limbic regions at baseline and change from baseline after metformin treatment
Time Frame: Baseline, 20 weeks, 40 weeks
Population: as for outcome 1
Arm/Group | Controls | Metformin | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Mu-opioid Receptor Binding Potential in Right Amygdala, Resting State
Description: Mu-opioid neurotransmission in limbic brain regions at baseline and change from baseline after metformin treatment
Time Frame: Baseline, 20 weeks, 40 weeks
Population: as for outcome 1
Arm/Group | Controls | Metformin | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Positive and Negative Affect Schedule - Positive Affective State
Description: Compare positive affective state between controls and insulin resistant women. Positive and Negative Affect Schedule - positive affective state. Scores can range from 10-50, with higher scores representing more positive affective state (better outcome)
Time Frame: Baseline
Population: All women assessed at baseline, prior to treatment arm randomization, so all insulin resistant women are analyzed as a single group. On the Control side, one woman's data for affective state is unavailable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controls | Insulin Resistant Participants
Number analyzed (Participants) | 26 | 12
units on a scale | 28.23 (8.29) | 21.83 (8.84)

6. Secondary Outcome: Positive and Negative Affect Schedule - Negative Affective State
Description: Measure of overall negative affective state at baseline in controls and insulin resistant women.
  Positive and Negative Affect Schedule - negative affective state. Scores can range from 10-50, with higher scores representing more negative affective state (worse outcome)
Time Frame: Baseline
Population: All women assessed at baseline, prior to treatment arm randomization, so all insulin resistant women analyzed as a single group. One woman's baseline affective score is not available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controls | Insulin Resistant Participants
Number analyzed (Participants) | 26 | 12
units on a scale | 11.46 (1.68) | 12.83 (6.74)

7. Secondary Outcome: Profile of Mood States - Overall Negative Mood
Description: Measure of overall negative mood at baseline in controls and insulin resistant women; Profile of Mood States are standardized to a relative score where a higher score is a worse mood state. Standardized cores generally ranged from - 11 to 52.
Time Frame: Baseline
Population: All women assessed at baseline, prior to treatment arm randomization, so all insulin resistant women analyzed as a single group; one woman on the control side's data is not available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controls | Insulin Resistant Participants
Number analyzed (Participants) | 26 | 12
units on a scale | 3.15 (10.60) | 14.42 (20.35)

8. Secondary Outcome: Beck Depression Index
Description: Measure of depression symptoms at baseline in controls and insulin resistant women. The Beck Depression Index runs on a scale from 0 to 63 where low scores mean less depression and high scores mean greater depression. Clinically, scores of 14 or higher are considered mild depression; 20 is moderate and 29 is severe.
Time Frame: Baseline
Population: All women assessed at baseline, prior to treatment arm randomization, so all insulin resistant women analyzed as a single group. The data for one woman in the control group is unavailable. Note: women with BDI scores of greater than 20 were excluded from the study by definition and therefore could not be in either arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Controls | Insulin Resistant Participants
Number analyzed (Participants) | 26 | 12
units on a scale | 2.93 (4.36) | 7.00 (9.96)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 40 weeks of study participation.
Groups:
- Placebo (First Assignment & Washout or Second Assignment): Placebo comparator to metformin treatment
  Placebo: Placebo capsules prepared identically to Metformin capsules
- Metformin (First Assignment & Washout or Second Assignment): 16 weeks treatment with metformin (insulin sensitizing treatment)
  Metformin: Women classified as insulin resistant will participate in both a placebo and a metformin treatment arm, each lasting about 16 weeks. Women will be randomized to order of treatment arms.
- Insulin-resistant Women Not Randomized: These participants, like controls, did not continue beyond baseline and were not assigned any metformin or placebo.
Arm/Group | Controls | Placebo (First Assignment & Washout or Second Assignment) | Metformin (First Assignment & Washout or Second Assignment) | Insulin-resistant Women Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/5 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/5 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 2/30 | 2/5 | 0/3 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Controls (N=30) | Placebo (First Assignment & Washout or Second Assignment) (N=5) | Metformin (First Assignment & Washout or Second Assignment) (N=3) | Insulin-resistant Women Not Randomized (N=6)
Nausea? (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated potassium levels (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Self-reported seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant reported undiagnosed seizure during placebo treatment; study participation was halted
Brain lesion detected (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Brain lesion was detected during study MRI scan. Participant notified and spoke with study radiologist, and referred to diagnostic radiologist care.

LIMITATIONS AND CAVEATS:
A limitation of this study is the relatively small sample size of the insulin resistant group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT02069379/Prot_SAP_000.pdf